CLINICAL TRIAL: NCT00177970
Title: Intravenous Immunoglobulin G Versus Placebo for the Treatment of Patients With Severe Clostridium Difficile-Associated Diarrhea and Colitis
Brief Title: IVIG Versus Placebo for the Treatment of Patients With Severe C-Diff
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We were unable to receive IVIG free from phamaceutical company.
Sponsor: University of Pittsburgh (Other)
Collaborators: Shadyside Hospital Foundation (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0311034
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Clostridium Difficile-associated Diarrhea (CDAD)
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG (Active Comparator)
  Interventions: Drug: intravenous immunoglobulin G (IVIG)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: intravenous immunoglobulin G (IVIG) — IVIG to be given IV to patients with C-Diff .
  Other Names: IVIG
  Arms: IVIG
Drug: Placebo — Placebo to be given IV to patients with C-Diff
  Arms: Placebo

SUMMARY:
In this trial, eligible patients will be randomly assigned to receive a single dose of 400 mg/kg of IVIG or a normal saline infusion as placebo over 4-6 hours, in addition to their usual medications for CDAD. We expect to enroll approximately 40 patients over a period of two years from UPMC Shadyside Hospital, McKeesport Hospital, and St. Margaret's Hospital who are unresponsive to standard antimicrobial therapy for CDAD.

During the course of this study we expect that IVIG group compared with placebo group will have fewer number of stools per day (< 3 per day). Secondary endpoints will include normal WBC count, normal body temperature, 75% reduction in abdominal pain / tenderness, and decrease in length of hospital stay.

Subjects will sign a written informed consent prior to any study procedures. Patients will be monitored closely during the infusion of the study medication and will continue to be monitored on a daily basis up to the time of discharge. Data collection will include vital signs, CBC, stool C. difficile cytotoxin assay, and stool counts before and after therapy.

DETAILED DESCRIPTION:
See "Brief Summary" for details

ELIGIBILITY:
Inclusion Criteria:

1. Males and female greater than 18 years of age
2. Positive stool C. difficile cytotoxin assay and/or biopsy evidence of Pseudomembranous Colitis (PMC) at onset of illness
3. Current history of severe, relapsing CDAD or Current history of severe, refractory CDAD
4. A score of 6 or 7 on the C.Diff Severity and Prognosis Score (CDSPS) scale27,28,29,30 OR failure to respond (as identified by a score of 4 or more on the CDSPS scale below) to any of the following: a 4-day or more course of oral or IV metronidazole 500 mg po TID or QID; or to a 4-day course of oral vancomycin 125-500 mg po Q6 hours; or to a 4-day course of vancomycin enemas; or failure to respond to a 4-day course of combination therapy of oral vancomycin 125-500 mg po Q6 hours and IV metronidazole 500mg IV Q8 or Q6 hours and/or vancomycin enemas.

CDSPS SCALE (each item is scored as one point for a 7 point maximum total)

1. underlying immunosuppression/chronic medical condition
2. altered or depressed mental status as defined by medical chart documentation
3. abdominal pain and/or distention
4. WBC > 20,000 or < 1,500 and/or bandemia > 10%
5. hypoalbuminemia (<3 mg/dL)
6. ascites (clinically or per CT scan findings per medical chart)
7. abnormal CT scan findings per medical chart -

Exclusion Criteria:

1. Pregnant or lactating women
2. Selective IgA deficiency
3. Hypersensitivity to immune globulin, human albumin, or thimerosal -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Arnold, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - UPMC McKeesport Hospital and SemperCare Hospital of McKeesport, Inc, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC St. Margaret Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
records not available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment number retrieved from old IRB database and not from study records and cannot be verified.
Period: Overall Study
Arm/Group | IVIG | Placebo
Started | 0 (No results available record destroyed due to age of study. no publications) | 0 (No results available record destroyed due to age of study. no publications)
Completed | 0 (No results available record destroyed due to age of study. no publications) | 0 (No results available record destroyed due to age of study. no publications)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No results available record destroyed due to age of study. no publications
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants] — No results available record destroyed due to age of study. no publications
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: 1) Normalization of WBC's
Description: During the course of the study, we expect the IVIG group compared to the placebo group will have a normal WBC count 3.8-10.0/CMM
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: 2) Decrease of Number of Loose Stools to <3 Per Day Following Treatment
Description: During the course of the study, we expect the IVIG group compared to the placebo group will have fewer number of stools per day (<3 per day).
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: 1) 75% Reduction in Abdominal Pain/Tenderness
Description: During the course of the study, we expect the IVIG group compared to the placebo group will a 75% reduction in abdominal pain/tenderness
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: 2) Quantity of Anti-C. Difficile Antibodies in Relationship With Recovery of C. Difficile Diarrhea
Description: The quantity of anti-C. difficile antibodies with improve in relationship with recovery
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 3) Correlation Between Antibody Responses as Measured With ELISA (Enzyme Immunoassay) and Recovery of C. Difficile Diarrhea
Description: A correlation will occur between antibody responses as measured with ELISA (enzyme immunoassay) and recovery of C. difficile diarrhea.
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: 4) Normalization of Neutrophil Count on CBC With Diff.
Description: During the course of the study, we expect the IVIG group compared to the placebo group will have normalization of neutrophil count (1.6-6.7)on CBC with diff.
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: 5) Normalization of Body Temperature During a 24 Hour Period
Description: During the course of the study, we expect the IVIG group compared to the placebo group will have a normal body temperature of 98.6 F.
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: 6) Patients' Length of Hospital Stay
Description: During the course of the study, we expect the IVIG group compared to the placebo group will have a decrease in length of hospital stay.
Time Frame: during the course of the study
Population: No results available record destroyed due to age of study. no publications
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No results available. Records were destroyed due to age of study.
Arm/Group | IVIG | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No